CLINICAL TRIAL: NCT03429270
Title: A Pivotal Study to Assess the Performance, Safety and Usability of a New 5 French Air-Charged Catheter for Performing Urodynamic Studies on Pediatric Subjects
Brief Title: T-DOC® 5 Fr Pediatric Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TDOC5Fr-PEDS-01-PR
Record Dates: First submitted 2018-01-19; First posted 2018-02-12 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Urodynamics Arm (Experimental)
  Interventions: Device: TDOC 5Fr

INTERVENTIONS:
Device: TDOC 5Fr — A Pivotal Study to Assess the Performance, Safety and Usability of a New 5 French Air-Charged Catheter for Performing Urodynamic Studies on Pediatric Subjects

SUMMARY:
A Pivotal Study to Assess the Performance, Safety and Usability of a New 5 French Air-Charged Catheter for Performing Urodynamic Studies on Pediatric Subjects

ELIGIBILITY:
Inclusion Criteria:

* Male and Female (Children and infants, 12 years of age and younger)
* Subjects who are scheduled and normally indicated for urodynamics testing, for any medically necessary reason as per the physician.

Exclusion Criteria:

* Subjects who suffer from bladder infections (not including subjects with asymptomatic bacteruria)
* Subjects with urethral strictures
* Subjects who require the use of a suprapubic catheter

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female and male pediatric
Enrollment: 28 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Virginia Health System - UVA - Pediatric Urology Clinic, Charlottesville, Virginia
  - J.W. Ruby Memorial Hospital and WVU Medicine Children's, Morgantown, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Urodynamics Arm: Urodynamic testing and data collection(per protocol) using the TDOC 5Fr catheters.
Period: Overall Study
Arm/Group | Urodynamics Arm
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in Which the T-DOC® 5 Fr Catheters Are Safe in Measuring Urodynamic Pressures in Pediatric Subjects (12 Years of Age and Younger).
Description: A binary clinician response after each UDS study is used to assess if it is clinically adequate (success) or inadequate (failure) in each patients questionnaire and presented to the clinician where safety (Yes the device is safe and No the device is not safe) will be reported. A minimum of 10 male and 10 female subjects, with an overall minimum of 28, and maximum of 33 subjects.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 28
Participants | 28

2. Primary Outcome: The Number of Patients in Which the T-DOC® 5 Fr Catheters Are Effective in Measuring Urodynamic Pressures in Pediatric Subjects (12 Years of Age and Younger).
Description: A binary clinician response after each UDS study is used to assess if it is clinically adequate (success) or inadequate (failure) in each patients questionnaire and presented to the clinician where effectiveness (Yes the device is effective and No the device is not effective) will be reported. A minimum of 10 male and 10 female subjects, with an overall minimum of 28, and maximum of 33 subjects.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 28
Participants | 28

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 to 7 days
Arm/Group | Urodynamics Arm
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urodynamics Arm (N=28)
Dysuria (Renal and urinary disorders) | 3 (3)
Hematochezia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03429270/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT03429270/SAP_001.pdf